CLINICAL TRIAL: NCT03471000
Title: The Influence of the Crown-implant Ratio on the Crestal Bone Level and Implant Secondary Stability - 36 Months Clinical Study
Brief Title: The Influence of the Crown-implant Ratio on the Crestal Bone Level and Implant Secondary Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Hadzik (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry); Wrocław Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Jakub Hadzik, PhD, DDS, Medical Innovation Center Wroclaw
Organization: Medical Innovation Center Wroclaw (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: crown-implant ratio
Record Dates: First submitted 2018-03-05; First posted 2018-03-20 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Partial Edentulism; Tooth Loss
Keywords: implant; dental implant
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short implants Treatment (Experimental): Group 2 (G2; n=15 patients) had short implants (OsseoSpeed ™ L6mm Ø4 mm) [DENTSPLY Implants, Waltham, MA, USA] placed without sinus lift and augmentation procedure.
  Interventions: Other: Short implants Treatment
- Regular Implants Treatment (Active Comparator): Group 1 (G1; n=15 patients) had conventional dental implants (OsseoSpeed ™ L11 Ø4 mm and L13 Ø4 mm) [DENTSPLY Implants, Waltham, MA, USA] placed, preceded by the sinus lift procedure from a lateral window approach with the application of the xenogeneic bone graft Geistlich Bio-Oss® [Geistlich AG, Wolhusen, Switzerland]. The lateral window approach sinus lift surgery was performed 6 weeks prior to the implant placement by the same surgeon.
  Interventions: Other: Regular implants Treatment

INTERVENTIONS:
Other: Short implants Treatment — Short implants are placed in the alveolar bone and a clinical Ostell and Periotest evaluation of the implants after a period of time is done. Analysis of periapical radiographs and CBCT images after a period of time. Bone around the implant was measured, marginal bone level loss is determined.
  Arms: Short implants Treatment
Other: Regular implants Treatment — Sinus lift procedure is done and regular implants are placed in the alveolar bone and a clinical Ostell and Periotest evaluation of the implants after a period of time is done. Analysis of periapical radiographs and CBCT images after a period of time. Bone around the implant was measured, marginal bone level loss is determined.
  Arms: Regular Implants Treatment

SUMMARY:
The aim of the study was to determine whether implant length and the crown-to-implant (C/I) ratio influence implant stability and the loss of the surrounding marginal bone, and whether short implants can be used instead of sinus augmentation procedures.

DETAILED DESCRIPTION:
The patients participating in the study (n=30) had one single tooth implant - a short (OsseoSpeed™ L6Ø4 mm, Implants) or a regular implant (OsseoSpeed™ L11 and L13Ø4 mm, DENTSPLY Implants) - placed in the maxilla. The evaluation was based on clinical and radiological examination.

The crown-to-implant ratio was determined by dividing the length of the crown together with the abutment by the length of the implant placed crestally. Mean crown-to-implant ratios were calculated separately for each group and its correlation with the MBL (marginal bone loss) and stability was assessed. The authors compared the correlation between the C/I ratio values, MBL and secondary implant stability.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking patients with no systemic or local diseases were qualified.

Additional inclusion criteria were as follows:

* minimal apicocoronal height of the alveolar ridge of 6 mm in the region of the implant insertion in the pre-surgical qualification
* minimal width of the alveolar ridge of 6-7 mm in the region of interest
* HKT (height of the keratinized tissue) higher than 2 mm
* API ≤ 35 (Approximal Plaque Index)
* PI ≤ 25. (Plaque Index)
* Bone Type III or D2 were included in the study
* No graft procedures in the area of interest,

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical measurement of implant stability | 36 months
  Evaluation of implant secondary stability in both groups. Stability measured and evaluated with Periotest(R) device - after 36 months.

SECONDARY OUTCOMES:
Radiological measurement of marginal bone loss around implant | 36 months
  Evalation if there is difference in marginal bone level around the implants in both groups. Periapical radiographs and CBCT images taken and the begining and at the end of the observation period will be compared and bone level will be measured. Loss of marginal bone will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Dominiak, Prof, Principal Investigator — Medical University Wrocław

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hadzik J, Krawiec M, Slawecki K, Kunert-Keil C, Dominiak M, Gedrange T. The Influence of the Crown-Implant Ratio on the Crestal Bone Level and Implant Secondary Stability: 36-Month Clinical Study. Biomed Res Int. 2018 May 16;2018:4246874. doi: 10.1155/2018/4246874. eCollection 2018. PMID 29862269